CLINICAL TRIAL: NCT00776594
Title: Randomized Phase II Trial of Short-Course Androgen Deprivation Therapy +/- Bevacizumab for PSA Recurrence of Prostate Cancer After Definitive Local Therapy
Brief Title: Androgen Deprivation Therapy +/- Bevacizumab for PSA Recurrence of Prostate Cancer After Definitive Local Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Associate Professor of Medicine, HMS, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-190; NCT01019031 (obsolete NCT alias)
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Prostate Cancer
Keywords: Androgen deprivation therapy; ADT; bevacizumab
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; bicalutamide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Androgen Deprivation Therapy Plus Bevacizumab
  Interventions: Drug: Androgen Deprivation Therapy; Drug: bicalutamide; Drug: bevacizumab
- Group 2 (Experimental): Androgen Deprivation Therapy Alone
  Interventions: Drug: Androgen Deprivation Therapy; Drug: bicalutamide

INTERVENTIONS:
Drug: Androgen Deprivation Therapy — leuprolide: 22.5mg given IM every 3 months for a total of 6 months or, goserelin acetate: 10.8mg given SC every 3 months for a total of 6 months
  Other Names: ADT
Drug: bicalutamide — 50mg orally daily for 6 months
Drug: bevacizumab — 15mg/ks given IV every three weeks for a total of 8 infusions over 6 months
  Arms: Group 1

SUMMARY:
The purpose of this research study is to assess the efficacy of antiangiogenic therapy (bevacizumab) and androgen deprivation versus androgen deprivation alone at the time of minimal systemic disease (based on rising PSA without metastases).

DETAILED DESCRIPTION:
* Participants will be randomized into one of two study groups. The first group will receive Androgen Deprivation Therapy (ADT) plus bevacizumab. The second group will receive ADT alone.
* For the Androgen Deprivation therapy either (treating physician discretion)leuprolide or goserelin acetate (given as injections) every 3 months for a total of 6 months. Bicalutamide will also be taken orally daily for a total of 6 months.
* Bevacizumab will be given intravenously every three weeks for a total of 8 infusions over 6 months.
* Participants will be evaluated every 7-9 weeks with vitals, physical exam, PS, laboratories including PSA and testosterone.

ELIGIBILITY:
Inclusion Criteria:

* History of biopsy documented prostate cancer (any Gleason score)
* Past treatment with prostatectomy with or without salvage prostate/pelvic radiation or primary radiation (external beam or brachytherapy)
* If past prostatectomy, pathologic stage no greater than T1-3, N1, M0
* PSA recurrence with PSAdt < 18 months. There is no minimum PSA for prostatectomy patients. For patients treated with primary radiation therapy PSA should be greater than 2.0 ng/ml
* No evidence of recurrent disease on exam, bone scan, CT/MRI abdomen/pelvis or CXR
* Prior ADT allowed if < 6 months and testosterone recovered to within 50 units (ng/dl) of normal range
* ECOG Performance status of 0-1
* Absolute neutrophil count of >1,500
* Platelet count > 100,000
* Hg > 8g/dl
* No history of bleeding or thromboses within the last 12 months that required medical intervention

Exclusion Criteria:

* History of cancer within 5 years, other than prostate cancer and non-melanoma skin cancer
* Medical condition requiring concomitant corticosteroids
* Active infection
* Prior chemotherapy allowed if was < 6 cycles and > 6 months prior to study entry
* Documented local recurrence or metastatic prostate cancer
* Inability to comply with study and/or follow-up procedures
* Life expectancy of less than 2 years
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-10; Primary Completion 2014-12 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Johns Hopkins University, Baltimore, Maryland
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The University of Texas M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Androgen Deprivation Therapy Plus Bevacizumab: Androgen Deprivation Therapy Plus Bevacizumab
  Androgen Deprivation Therapy: leuprolide: 22.5mg given IM every 3 months for a total of 6 months or, goserelin acetate: 10.8mg given SC every 3 months for a total of 6 months
  bicalutamide: 50mg orally daily for 6 months
  bevacizumab: 15mg/ks given IV every three weeks for a total of 8 infusions over 6 months
- Androgen Deprivation Therapy Alone: Androgen Deprivation Therapy Alone
  Androgen Deprivation Therapy: leuprolide: 22.5mg given IM every 3 months for a total of 6 months or, goserelin acetate: 10.8mg given SC every 3 months for a total of 6 months
  bicalutamide: 50mg orally daily for 6 months
Period: Overall Study
Arm/Group | Androgen Deprivation Therapy Plus Bevacizumab | Androgen Deprivation Therapy Alone
Started | 66 | 36
Completed | 62 | 34
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgen Deprivation Therapy Plus Bevacizumab | Androgen Deprivation Therapy Alone | Total
Number analyzed (Participants) | 66 | 36 | 102
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [60 to 69] | 63 [60 to 68] | 65 [65 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 66 | 36 | 102

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival
Description: To identify a difference in relapse-free survival in men treated with short course ADT (6 months) versus short course ADT plus bevacizumab.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 66 | 36
months | 13 [11 to 15] | 10 [10 to 12]

2. Secondary Outcome: Number of Participants With PSA <0.2 ng/ml at Six Months
Description: Number of participants with a PSA <0.2 ng/ml at six months (upon completion of treatment).
Time Frame: Six months (at completion of treatment)
Measure: Number; unit: Number of participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 64 | 35
Number of participants | 51 | 27

3. Secondary Outcome: Cardiovascular Safety Including Measurement of Blood Pressure During Treatment Period (6 Months).
Description: The number of patients who developed hypertension (greater that 150 systolic or greater than 90 diastolic) during treatment period.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 65 | 36
participants | 48 | 13

4. Secondary Outcome: Analysis of Cytokines and Angiogenic Factors in Plasma/Serum
Description: Analysis of cytokines and angiogenic factors in plasma/serum at baseline and at 6 months (end of treatment).
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Leptin Level in Patients Treated With ADT+Bev: Leptin level in patients with sample available treated with ADT+bev
- Leptin in Patients Treated With ADT Alone: Leptin in patients with sample available treated with ADT alone
Arm/Group | Leptin Level in Patients Treated With ADT+Bev | Leptin in Patients Treated With ADT Alone
Number analyzed (Participants) | 43 | 21
pg/ml | 13755 [6570 to 25762] | 10179 [6924 to 15333]

ADVERSE EVENTS:
Arm/Group | Group 2 | Group 1
Serious Adverse Events (participants affected / at risk) | 5/36 | 18/66
Other Adverse Events (participants affected / at risk) | 32/36 | 63/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 2 (N=36) | Group 1 (N=66)
Cardiac-ischemia (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 13
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Infection w/ unk ANC peritoneal cavity (Infections and infestations) | 0 | 1
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Head/headache (Nervous system disorders) | 0 | 1
Bronchospasm- wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 2 (N=36) | Group 1 (N=66)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Allergy-other (Immune system disorders) | 0 | 1
Bone marrow cellularity (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 3 | 3
Leukocytes (Investigations) | 1 | 0
Lymphopenia (Investigations) | 0 | 2
Platelets (Investigations) | 0 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 1
Arrhythmia-other (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 19
Fatigue (General disorders) | 8 | 38
Fever w/o neutropenia (General disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 7
Rigors/chills (General disorders) | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 2 | 3
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 2
Constitutional- other (General disorders) | 0 | 3
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 1 | 5
Hot flashes (Vascular disorders) | 25 | 42
Hyopthyroidism (Endocrine disorders) | 0 | 1
Endocrine-other (Endocrine disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 9
Dentures or dental prosthesis (Gastrointestinal disorders) | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Fistula- Anus (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Incontinence- anal (Gastrointestinal disorders) | 1 | 1
Muco/stomatitis by exam- larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 0 | 2
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 2
Muco/stomatitis (symptom) stomach (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Salivary (Gastrointestinal disorders) | 0 | 1
Taste disturbance (Nervous system disorders) | 0 | 2
Ulcer- duodenum (Gastrointestinal disorders) | 0 | 1
GI-other (Gastrointestinal disorders) | 1 | 2
Lower GI- hemorrhage NOS (Gastrointestinal disorders) | 2 | 2
Oral cavity- hemorrhage (Gastrointestinal disorders) | 0 | 4
Rectum- hemorrhage (Gastrointestinal disorders) | 0 | 1
Bladder- hemorrhage (Renal and urinary disorders) | 0 | 1
Urinary hemorrhage NOS (Renal and urinary disorders) | 1 | 2
Nose- hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 15
Hemorrhage-other (Vascular disorders) | 0 | 1
Infection Gr0-2 neut- bronchus (Infections and infestations) | 0 | 1
Infection Gr0-2 neut- oral cavity (Infections and infestations) | 0 | 1
Infection Gr0-2 neut- sinus (Infections and infestations) | 0 | 2
Infection Gr0-2 neut- upper airway (Infections and infestations) | 0 | 1
Infection Gr0-2 neut- urinary tract (Infections and infestations) | 0 | 1
Infection w/ unk ANC oral cavity/gums (Infections and infestations) | 0 | 1
Infection w/ unk ANC sinus (Infections and infestations) | 0 | 1
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 0 | 1
Infection-other (Infections and infestations) | 0 | 2
Edema head and neck (General disorders) | 0 | 1
Edema limb (General disorders) | 2 | 4
Lymphatics-other (Blood and lymphatic system disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Alkaline phosphatase (Investigations) | 0 | 1
ALT- SGPT (Investigations) | 2 | 4
AST- SGOT (Investigations) | 2 | 5
Bilirubin (Investigations) | 0 | 1
Hypercholesterolemia (Investigations) | 1 | 4
Creatinine (Investigations) | 0 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hemoglobinuria (Renal and urinary disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 7
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 4
Extremity-lower (gait/walking) (General disorders) | 1 | 0
Extremity upper (function) (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint-function (Musculoskeletal and connective tissue disorders) | 0 | 2
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 1
Nonneuropathic upper extr muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 2
Confusion (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 5
Memory impairment (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 2
Neuropathy CN II vision (Eye disorders) | 0 | 1
Neuropathy CN IX pharynx ear tongue (Nervous system disorders) | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 11
Neurologic-other (Nervous system disorders) | 0 | 2
Glaucoma (Eye disorders) | 1 | 0
Vision-blurred (Eye disorders) | 0 | 1
Ocular-other (Eye disorders) | 1 | 1
Abdomen- pain (Gastrointestinal disorders) | 0 | 2
Anus- pain (Gastrointestinal disorders) | 0 | 1
Back- pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Buttock- pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall- pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest/thoracic pain NOS (General disorders) | 0 | 2
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 1 | 9
Head/headache (Nervous system disorders) | 2 | 28
Joint- pain (Musculoskeletal and connective tissue disorders) | 2 | 15
Muscle- pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Neck- pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neuropathic- pain (Nervous system disorders) | 0 | 1
Oral cavity- pain (Gastrointestinal disorders) | 0 | 1
Scalp- pain (Skin and subcutaneous tissue disorders) | 0 | 1
Scrotum- pain (Reproductive system and breast disorders) | 0 | 1
Throat/pharynx/larynx- pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain-other (General disorders) | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstruction- airway-bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Incontinence urinary (Renal and urinary disorders) | 1 | 3
Urinary frequency/urgency (Renal and urinary disorders) | 4 | 15
Urinary retention (Renal and urinary disorders) | 0 | 1
Renal/GU-other (Renal and urinary disorders) | 1 | 2
Intra-op injury Face NOS (Injury, poisoning and procedural complications) | 0 | 1
Erectile impotence (Reproductive system and breast disorders) | 0 | 1
Libido (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No